CLINICAL TRIAL: NCT01758783
Title: the Efficacy of Glutamine in the Therapy of Radiation Enteritis Among Patients Treated With Radiation of Abdomen and Pelvis.
Brief Title: Therapy of Radiation Enteritis With Glutamine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Nanjing University School of Medicine (Other)
Responsible Party: Principal Investigator, Lei Zheng, Resident, Nanjing University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Radiation Enteritis 001
Record Dates: First submitted 2012-12-27; First posted 2013-01-01 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Radiation Enteritis
MeSH Terms: interventions — Glutamine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo group (Placebo Comparator)
  Interventions: Drug: Glutamine
- Glutamine group (Experimental)
  Interventions: Drug: Glutamine

INTERVENTIONS:
Drug: Glutamine — amino acid：1.2-2g/(kg·d) Glutamine：0.5g /(kg·d)

SUMMARY:
Objective: To evaluate the effects of perioperative glutamine supplemented total parenteral nutrition support on nutritional status, immunologic function and intestinal permeability of patients with chronic radiation intestinal injury.

Methods: The 40 patients with CRII were randomized into two groups, the standard TPN group and glutamine-enriched TPN group. The patients were administered total parenteral nutrition for at least four weeks (two weeks pre-operation and two weeks post-operation). The nutritional status, immunologic function, plasma concentration of glutamine and intestinal permeability were measured at 1 day, 1 week and 2 weeks pre-operation, 3 day, 1 week and 2 weeks post-operation. Nutrition status was determined the plasma concentrations of hemoglobin, albumin, prealbumin, transferrin and triglyceride. Immunologic function were measured by the percentages of CD4+T cells and CD8+T cells, the ratio of CD4 +T cells to CD8+T cells ( CD4 +/CD8 +) was calculated， and serum IgA, IgM and IgG．The intestinal permeability was detected by the urinal ratio of lactulose and mannitol.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic radiation enteritis
* Need the operation
* Malnutrition

Exclusion Criteria:

* Hepatic failure
* Kidney failure
* Neoplasm recurrence
* Serious cardiovascular/metabolic disease
* Pregnancy and lactation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-06 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
inflammatory factor | 2 weeks after the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Nanjing General Hospital of Nanjing Command, Nanjing, Jiangsu, China